CLINICAL TRIAL: NCT02343302
Title: Prospective Trial Evaluating the Effect of Closed Suction Drainage Versus Straight Drainage After Distal Pancreatectomy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor patient accrual
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NA_00080937; IRB00197557 (Other: Johns Hopkins IRB)
Record Dates: First submitted 2015-01-15; First posted 2015-01-21 (Estimated); Results first posted 2021-12-21 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-03

CONDITIONS: Pancreatic Fistula
Keywords: Pancreatic Fistula
MeSH Terms: conditions — Pancreatic Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Soft Pancreatic Gland (Other): This arm will be patients with glands felt to have a soft texture during surgery. This arm will receive either a suction drain or a gravity drain based on the note inside the sealed envelope.
  Interventions: Device: Jackson-Pratt Drain; Device: Non-suctioning drainage
- Hard Pancreatic Gland (Other): This arm will include patients felt to have a hard gland tecture at the time of surgery. This arm will receive either a suction drain or a gravity drain based on the note inside the sealed envelope.
  Interventions: Device: Jackson-Pratt Drain; Device: Non-suctioning drainage

INTERVENTIONS:
Device: Jackson-Pratt Drain — A closed suctioning drain will be placed at the time of surgery. Patients in both arm A and arm B will receive this intervention. The patients that receive this treatment will be the ones whose envelope, selected on the basis of the texture of the gland, contains a card labelled "suction drain"
Device: Non-suctioning drainage — A closed non-suctioning drain will be placed at the time of surgery. Patients in both arm A and arm B will receive this intervention. The patients that receive this treatment will be the ones whose envelope, selected on the basis of the texture of the gland, contains a card labelled "gravity drain"

SUMMARY:
A very common complication following distal pancreatectomy is leakage from the pancreas, or what is called a pancreatic fistula. We hypothesize that operative drains which create suction may contribute to the development of leakage from the pancreas. This study evaluates the effect of using non-suctioning drains to prevent the development of this complication.

DETAILED DESCRIPTION:
The most common complication following distal pancreatectomy is the developement of leakage from the remaining pancreas gland, which results in significant morbidity. Most surgeons leave dains at the time of surgery to prevent complications from pancreatic leakage. However, we hypothesize that drains which create continous negative pressure may contribute to the development of a pancreatic fistula. This study randomizes patients to suctioning versus non-suctioning drains. The primary endpoint is the development of pancreatic fistuale, as defined by the International Study Group of Pancreatic Surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing distal pancreatectomy at Johns Hopkins Hospital

Exclusion Criteria:

* Children <18 years old, pregnant women, adults lacking capacity to consent, non-english speakers, and prisoners.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher L Wolfgang, MD PHD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Soft Pancreatic Gland | Hard Pancreatic Gland
Started | 1 | 1
Completed | 0 | 0
Not Completed | 1 | 1
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Population: Work on this project was discontinued. Baseline data was not collected for any participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Soft Pancreatic Gland | Hard Pancreatic Gland | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Pancreatic Fistula
Description: The primary endpoint of the study is the developement of post-operative pancreatic fistula, as defined by the International Study Group of Pancreatic Surgery.
Time Frame: 90 days
Population: Work on this project was discontinued due to poor recruitmemt. Data was not collected for this outcome measure.
Arm/Group | Soft Pancreatic Gland | Hard Pancreatic Gland
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Morbidity
Description: All morbidity, including length of hospital stay, need for enteral/parenteral nutrition, need for radiologic/surgical intervention, septic complications, and peri-operative mortality.
Time Frame: 90 days
Population: Work on this project was discontinued due to poor recruitmemt. Data was not collected for this outcome measure.
Arm/Group | Soft Pancreatic Gland | Hard Pancreatic Gland
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Not applicable. Work on this project was discontinued. No adverse event data was collected.
Description: No adverse event data was collected.
Arm/Group | Soft Pancreatic Gland | Hard Pancreatic Gland
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2012-12-08): https://cdn.clinicaltrials.gov/large-docs/02/NCT02343302/Prot_SAP_000.pdf
  • Informed Consent Form (2013-01-22): https://cdn.clinicaltrials.gov/large-docs/02/NCT02343302/ICF_001.pdf